CLINICAL TRIAL: NCT04507113
Title: Prognostic Value Assessment of Biomarkers in Acute Lumbar Radiculalgia : Contribution of the Diffusion Tensor in Magnetic Resonance Imaging
Brief Title: Diffusion Tensor (DTI) for the Assessement of Therapeutic Evolution of Patients With Acute Lumbar Radiculalgia
Acronym: DiTi-Aïe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0074
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Radiculopathy; Magnetic Resonance Imaging; Diffusion Tensor Imaging
Keywords: Lumbar Radiculopathy; Magnetic Resonance Imaging; Diffusion Tensor Imaging; Prognostic
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbar radiculopathy (Experimental): Patients with acute lumbar radiculopathy (less than 3 months of evolution)
  Interventions: Other: DTI sequence acquisition

INTERVENTIONS:
Other: DTI sequence acquisition — DTI sequence acquisition

SUMMARY:
Diffusion tensor imaging (DTI) is a non-invasive MRI technique offering a functional approach that provides morphological information about the microstructures of the nerve roots. DTI is a widely used neuroimaging technique and is a current topic of research in the field of peripheral nerve imaging.The aim of the study is to determine the prognostic quality of the DTI parameters to predict the therapeutic evolution of patients with lumbar radiculalgia at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Patient with Lumbar Radiculalgia (L4, L5 or S1)
* Pain VAS (Visual analog scale) > 30/100
* Less than 3 months of evolution
* With a radiculalgia superior or equal to lumbalgia
* Disco radicular conflict, verified by MRI
* Able to receive information
* Affiliated to French social security

Exclusion Criteria:

* History of chronic lumbalgia and radiculalgia
* History of lumbar surgery
* Recent episode (less than 6 months) with the same radicular topography
* Bilateral radicular compression on MRI
* Patient requiring emergency surgery
* Evolutive disease interfering with pain assesment (neoplasia, inflammatory rheumatism, peripheral neuropathy, central neurological disease)
* MRI contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-10-06 (Estimated); Study Completion 2025-11-06 (Estimated)

PRIMARY OUTCOMES:
Predictive performance of DTI imaging on the therapeutic evolution | 6 months
  DTI is a sensitive probe of cellular structure that works by measuring the diffusion of water molecules. The measured quantity is the diffusion coefficient, a proportionality constant that relates diffusive flux to a concentration gradient and has units of mm2/s.
  The objective is to know if the interpretation of DTI allow to predict the therapeutic evolution of patients. For instance, the patients will need in the future oral drugs? Or they will need rather an infiltration? Or they will need rather a surgery?

SECONDARY OUTCOMES:
Correlation between DTI parameters and pain intensity | 6 months
  DTI is a sensitive probe of cellular structure that works by measuring the diffusion of water molecules. The measured quantity is the diffusion coefficient, a proportionality constant that relates diffusive flux to a concentration gradient and has units of mm2/s.
  The intensity of pain will be self evaluated by the visual analogue scale (VAS). This scale is between 0 and 10 (in cms) being absence of pain and 10 intolerable pain.
Correlation between DTI parameters evolution and neuropathic pain | 6 months
  DTI is a sensitive probe of cellular structure that works by measuring the diffusion of water molecules. The measured quantity is the diffusion coefficient, a proportionality constant that relates diffusive flux to a concentration gradient and has units of mm2/s.
  The presence of neuropathic pain will be evaluated by the Neuropathic Pain Symptom Inventory (NPSI) scale. This is a self-questionnaire.The tool evaluates mean pain intensity in the last 24h in a verbal numeric scale from zero (no pain) to 10 (worst imaginable pain). Total pain intensity score may be calculated by the sum of 10 descriptors.
Correlation between DTI parameters evolution and disability | 6 months
  DTI is a sensitive probe of cellular structure that works by measuring the diffusion of water molecules. The measured quantity is a diffusion coefficient, a proportionality constant that relates diffusive flux to a concentration gradient and has units of mm2/s. The disability will be measured by the Oswestry Disability Index (ODI). The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François BUDZIK, MD, PhD, Principal Investigator — Lille CU
Locations (1):
- Groupe Hospitalier de l'Institut Catholique de Lille, Lomme, France

IPD SHARING:
Plan to Share IPD: No